CLINICAL TRIAL: NCT02487199
Title: An Open-Label Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir With or Without Dasabuvir in Adults With Genotype 1a or Genotype 4 Chronic Hepatitis C Virus (HCV) Infection, With Severe Renal Impairment or End-Stage Renal Disease (RUBY-II)
Brief Title: Ombitasvir/Paritaprevir/Ritonavir With or Without Dasabuvir in Adults With Genotype 1a or Genotype 4 Chronic Hepatitis C Virus (HCV) Infection, With Severe Kidney Impairment or End Stage Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-461; 2015-002012-33 (EudraCT Number)
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: hepatitis C infection; hepatitis C; severe kidney disease; chronic kidney disease; Genotype 1a; Genotype 4; treatment experienced; interferon; IFN; pegIFN
MeSH Terms: conditions — Hepatitis C; Kidney Diseases; Renal Insufficiency, Chronic | interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCV GT1a (3-DAA) (Experimental): Participants with hepatitis C virus (HCV) genotype 1a (GT1a) infection received 3-direct-acting antiviral agent (3-DAA: ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir
- HCV GT4 (2-DAA) (Experimental): Participants with hepatitis C virus (HCV) genotype 4 (GT4) infection received 2-direct-acting antiviral agent (2-DAA: ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily]) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir, dasabuvir tablet
  Other Names: Viekira Pak, paritaprevir also known as ABT-450, ombitasvir also known as ABT-267, dasabuvir also known as ABT-333
  Arms: HCV GT1a (3-DAA)
Drug: ombitasvir/paritaprevir/ritonavir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir
  Other Names: Technivie, paritaprevir also known as ABT-450, ombitasvir also known as ABT-267
  Arms: HCV GT4 (2-DAA)

SUMMARY:
This study evaluates the efficacy and safety of ombitasvir/paritaprevir/ritonavir with or without dasabuvir in adults with hepatitis C virus (HCV) genotype 1a (GT1a) or genotype 4 (GT4) infection and with severe kidney impairment or end-stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus (HCV) genotype 1a (GT1a) infection or genotype 4 (GT4) infection (HCV RNA level greater than 1,000 IU/mL at Screening).
* Females must be post-menopausal, of non-child bearing potential or practicing specific forms of birth control.
* Chronic kidney disease stage 4 or stage 5.

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab)
* HCV genotype performed during screening unable to genotype or co-infection with any other HCV genotype, no mixed genotypes.
* Abnormal laboratory tests
* Current enrollment in another investigational study
* Prior treatment with a direct acting antiviral agent (DAA) containing regimen with the exception of interferon or pegylated interferon with or without ribavirin
* Current treatment with a direct acting antiviral agent (DAA) containing regimen
* Any evidence of liver cirrhosis or liver cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Derived] Shuster DL, Menon RM, Ding B, Khatri A, Li H, Cohen E, Jewett M, Cohen DE, Zha J. Effects of chronic kidney disease stage 4, end-stage renal disease, or dialysis on the plasma concentrations of ombitasvir, paritaprevir, ritonavir, and dasabuvir in patients with chronic HCV infection: pharmacokinetic analysis of the phase 3 RUBY-I and RUBY-II trials. Eur J Clin Pharmacol. 2019 Feb;75(2):207-216. doi: 10.1007/s00228-018-2566-6. Epub 2018 Oct 5. PMID 30291369
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 42-day screening period.
Period: Overall Study
Arm/Group | HCV GT1a (3-DAA) | HCV GT4 (2-DAA)
Started | 13 | 5
Completed | 13 | 4
Not Completed | 0 | 1
Not completed — Withdrew Consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCV GT1a (3-DAA) | HCV GT4 (2-DAA) | Total
Number analyzed (Participants) | 13 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.00) | 53.6 (14.08) | 54.5 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (<LLOQ) 12 weeks after the last dose of study drug. Participants with missing data after backward imputation were imputed as nonresponders.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCV GT1a (3-DAA) | HCV GT4 (2-DAA)
Number analyzed (Participants) | 13 | 5
percentage of participants | 100 [77.2 to 100.0] | 80.0 [37.6 to 96.4]

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity from first dose of study drug until 30 days after the last dose. For more details on AEs please see the Adverse Event section.
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks)
Population: Safety population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | HCV GT1a (3-DAA) | HCV GT4 (2-DAA)
Number analyzed (Participants) | 13 | 5
Participants
  Any TEAE | 13 | 5
  Any TESAE | 3 | 1

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment or confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment with at least 6 weeks of treatment.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCV GT1a (3-DAA) | HCV GT4 (2-DAA)
Number analyzed (Participants) | 13 | 5
percentage of participants | 0.0 [0.0 to 22.8] | 0.0 [0.0 to 43.4]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCV GT1a (3-DAA) | HCV GT4 (2-DAA)
Number analyzed (Participants) | 13 | 4
percentage of participants | 0.0 [0.0 to 22.8] | 0.0 [0.0 to 49.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any adverse event or serious adverse event that begins or worsens in severity after initiation of study drug until 30 days after the last dose of study drug.
Arm/Group | HCV GT1a (3-DAA) | HCV GT4 (2-DAA)
Serious Adverse Events (participants affected / at risk) | 3/13 | 1/5
Other Adverse Events (participants affected / at risk) | 13/13 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCV GT1a (3-DAA) (N=13) | HCV GT4 (2-DAA) (N=5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
FOLLICULITIS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
END STAGE RENAL DISEASE (Renal and urinary disorders) | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HCV GT1a (3-DAA) (N=13) | HCV GT4 (2-DAA) (N=5)
PALPITATIONS (Cardiac disorders) | 1 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 0
CUSHING'S SYNDROME (Endocrine disorders) | 1 | 0
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 1
DRY EYE (Eye disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 0
FLATULENCE (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 0
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0
ASTHENIA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 0
FATIGUE (General disorders) | 3 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1
PAIN (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
KIDNEY INFECTION (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
TRANSAMINASES INCREASED (Investigations) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
BURNING SENSATION (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 3 | 0
SCIATICA (Nervous system disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
EUPHORIC MOOD (Psychiatric disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 2 | 0
SLEEP DISORDER (Psychiatric disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 2 | 1
HYPOTENSION (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.